CLINICAL TRIAL: NCT03733613
Title: To Verify the Reliability and Validity of Kinect Detector While Apply to Physical Fitness Tests and Gait Performance Analysis
Brief Title: Reliability and Validity of Kinect Detector for Fitness Tests and Gait Performance Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM106054E
Record Dates: First submitted 2018-10-31; First posted 2018-11-07 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Healthy Adults
Keywords: Kinect; somatosensory detector; physical fitness; gait analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Subjects will receive pre and post-test, in order to verify the test-retest reliability of the Somatosensory detector
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Background: Depending on nature and needs, physical fitness can be divided into healthy fitness and physical fitness (also known as competitive fitness). Healthy fitness includes cardio-respiratory fitness, muscle fitness, muscular endurance, flexibility, and body composition. Physical fitness includes coordination, speed, explosiveness, balance, agility, and reaction time. Although the monitoring of fitness is very important, most of the tests need to be assisted by professionally trained fitness inspectors, so that the public who wants to regularly check their fitness status will facing a dilemma-- insufficient of inspectors. In the face of such a situation, the somatosensory detector may be a choice which is relatively objective, convenient and no need to rely on the inspectors. Therefore, the validity and retest reliability of the somatosensory detector need to be verified in order to achieve accurate and objective measurement results.

DETAILED DESCRIPTION:
Background: Depending on nature and needs, physical fitness can be divided into healthy fitness and physical fitness (also known as competitive fitness). Healthy fitness includes cardio-respiratory fitness, muscle fitness, muscular endurance, flexibility, and body composition. Physical fitness includes coordination, speed, explosiveness, balance, agility, and reaction time. Although the monitoring of fitness is very important, most of the tests need to be assisted by professionally trained fitness inspectors, so that the public who wants to regularly check their fitness status will facing a dilemma-- insufficient of inspectors. In the face of such a situation, the somatosensory detector may be a choice which is relatively objective, convenient and no need to rely on the inspectors. Therefore, the validity and retest reliability of the somatosensory detector need to be verified in order to achieve accurate and objective measurement results.

Research purposes: To verify the retest reliability and validity of the somatosensory detector on physical fitness and gait performance.

Methods: The trial will enroll 60 subjects, 30 of them were healthy individuals between the ages of 20 and 65, and 30 are healthy elderly than 65 years of age. The exclusion criteria including: (1) those who are unable to follow the instructions and who have orthopedic, nervous system or cardiopulmonary system disorders, or who have abnormal gait pattern, or who are affected by the above physiological system disorders. Subjects will receive two tests, there's a one-week interval between each test. In the first test, the fitness assessment of the fitness inspector and the somatosensory detector was performed simultaneously, and the fitness evaluation of the somatosensory detector was performed only for the second time. And use statistical software to analyze the reliability and validity of the somatosensory detector.

Statistical Analysis: Using SPSS 20.0 for data archiving and statistical analysis, the reliability and validity of the test will be detected by intraclass correlation one-way random model, and presenting by the intraclass correlation coefficient and 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* those unable to follow to instructions
* those have abnormal gait pattern which caused by orthopedics system disorders, nervous system disorders or cardio-respiratory disorders
* those with abnormal movement performance which caused by physiological system obstacles

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Change from baseline at one week
  Gait speed is calculated using distance in meters and time in seconds.
Gait cadence | Change from baseline at one week
  Cadence is the rate at which a person walk, expressed in steps per minute.
Gait stride length | Change from baseline at one week
  The stride length is the distance between two successive placements of the same foot.

SECONDARY OUTCOMES:
One leg standing test | Change from baseline at one week
  To test balance ability
Functional forward reach test | Change from baseline at one week
  To test functional balance performance
Timed up and go test | Change from baseline at one week
  To test functional balance performance
Upper arm curl test | Change from baseline at one week
  To test functional muscle strength of upper extremities
30 seconds sit-stand-sit test | Change from baseline at one week
  To test functional muscle strength of lower extremities
2 minutes stepping test | Change from baseline at one week
  To test cardiopulmonary ability

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan